CLINICAL TRIAL: NCT02307071
Title: Transcutaneous Suboccipital Neurostimulation for the Treatment of Chronic Migraine
Brief Title: Occipital Transcutaneous Stimulation in Chronic Migraine
Acronym: OSCRO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean Schoenen, Honorary Full Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTSCM
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cefaly Kit Arnold (Experimental): Occipital transcranial stimulation is implemented in occipital region at 16 mA of intensity, for 20 minutes, everyday for 3 months, in 20 chronic migraine patients.
  Interventions: Device: Cefaly Kit Arnold

INTERVENTIONS:
Device: Cefaly Kit Arnold — Occipital neurostimulation can have a therapeutic effect in chronic migraine treatment, thus representing a possible therapeutic option in patients that do not respond to any medication.

SUMMARY:
This study evaluates the effect in chronic migraine patients of daily 20 minute-transcutaneous sub occipital neurostimulation using the occipital Cefaly° device.

DETAILED DESCRIPTION:
Chronic migraine is a disabling neurological condition affecting 0.5-2% of the population.

CM is difficult to treat and preventive treatment options are limited. Due to the inefficiency of available and the lack of new preventive anti-migraine drug, neurostimulation methods have raised great interest in recent years.

The ONSTIM study showed a reduction in headache frequency in 39% of patients treated with active ONS during 12 weeks, compared to no improvement in the "non-effectively" stimulated or medically treated groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic migraine (ICHD III beta 1.3) with or without medication overuse

Exclusion Criteria:

* other diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Monthly frequency of migraine days | 2 months treatment

SECONDARY OUTCOMES:
Monthly frequency of headache days | 2 months
Monthly frequency of total headache days | 2 months
Cumulative monthly headache hours | 2 months
Monthly acute drug intake | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Schoenen, MD, PhD, Principal Investigator — University of Liege; Delphine Magis, MD, PhD, Principal Investigator — University of Liege
Locations (1):
- CHR Citadelle, Liège, Belgium, Belgium